CLINICAL TRIAL: NCT03641963
Title: Non-invasive Absolute Intracranial Pressure Measurement in Patients With Malignant Middle Cerebral Artery Infarction for Determination of Timing to Decompressive Craniectomy
Brief Title: aICP Measurement in Patients With Cerebral Artery Infarction / aICP MCA Infarction
Acronym: aICPStroke
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety questions on patients with glaucoma are in discussion by our IRB
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Javier Fandino, MD, Prof., Kantonsspital Aarau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: aICP Stroke
Record Dates: First submitted 2018-08-07; First posted 2018-08-22 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke patients with ICP measurement (Experimental): All patients with the possibility to evolve a malignant MCA infarct according to the initial assessment, will be included in our study, to measure ICP non-invasive. The ICP will be measured non-invasive with the Vittamed 205 Non-invasive intracranial pressure (ICP) meter.
  Interventions: Device: Vittamed 205 Non-invasive intracranial pressure (ICP) meter

INTERVENTIONS:
Device: Vittamed 205 Non-invasive intracranial pressure (ICP) meter — Non-Invasive intracranial pressure measurement

SUMMARY:
Space-occupying, malignant middle cerebral artery (M-MCA) infarctions are still one of the most devastating forms of ischemic stroke, with a mortality of up to 80% in untreated patients. It is reported that early hemicraniectomy leads to a substantial decrease in mortality at 6 and 12 months and is likely to improve functional outcome. Thus, this study investigates if non-invasive intracranial pressure (ICP) measuring could represent an objective value to determine the time point to indicate decompressive craniectomy surgery.

However, there are still important questions about the individual indication for decompressive surgery. In consideration of a variable clinical course (some patients develop fatal brain edema early, whereas other patients do not show severe brain swelling for several days), achieving a way to measure, control and predict malignant brain edema formation would be of extremely important value.

DETAILED DESCRIPTION:
Space-occupying, malignant middle cerebral artery (M-MCA) infarctions are still one of the most devastating forms of ischemic stroke, with a mortality of up to 80% in untreated patients.

Actually, M-MCA infarctions constitute between 1% to 10% of all supratentorial ischemic strokes, with a yearly incidence about 10-20/100.000 people. The etiology of malignant MCA infarctions is mostly due to thrombosis or embolic occlusion of either the internal carotid artery or the proximal MCA. The term M-MCA is referred to a severe MCA syndrome with typical clinical symptoms (hemiparesis to hemiplegia, severe sensory deficits, head and eye deviation, hemi-inattention, and, if the dominant hemisphere is involved, global aphasia), following a uniform clinical course (progressive deterioration of conscious within the first 24-48 h), and ending in herniation. An early diagnosis is essential and depends on CT (Computed Tomography) and MRI (Magnetic Resonance Imaging) to aid the prediction of a malignant course, but, until today there is no clear consensus to define and predict radiologically a malignant evolution in early phases.

Several pharmacological strategies have been proposed but the efficacy of these approaches has not been supported by adequate evidence from clinical trials and, until recently, treatment of malignant MCA infarctions has been a major unmet need.

Over the past 10 years, results from randomised controlled trials (RCT) (HAMLET, DECIMAL and DESTINY) and their pooled analyses have provided evidence that an early hemicraniectomy leads to a substantial decrease in mortality at 6 and 12 months and is likely to improve functional outcome. However, there are still important questions about the individual indication for decompressive surgery. In consideration of a variable clinical course (some patients develop fatal brain edema early, whereas other patients do not show severe brain swelling for several days), achieving a way to measure, control and predict malignant brain edema formation would be of extremely important value.

In this way, the ICP measuring could represent an objective value to determine in every patient the time point to indicate decompressive craniectomy surgery, and also could allow us to find a correlation between the size of the infarction and periinfarction edema. Therefore the optimal timing of surgical intervention can be defined and all the medical treatment adjusted.

Currently, ICP can be measured and registered only using invasive techniques. The two ICP measurement methods available - intraventricular and intraparenchymal - require both a neurosurgical procedure, in order to implant the catheter and probes within the brain. Thus, these measures include themselves a risk for the subject, and both infections and intracranial bleedings are regular albeit not frequent complications. In addition, invasive recording of ICP requires neurosurgical expertise and intensive care unit (ICU) facilities. Therefore ICP measurement so far, is not a standard of care in stroke units.

A reliable, accurate and precise non-invasive method to measure ICP would be of considerable clinical value, enabling ICP measurement without neurosurgical expertise and ICU facilities. Moreover, it would save the patients from the complication risks associated with invasive measures.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an ischemic stroke in the internal carotid artery or middle cerebral artery territory at risk of a malignant MCA evolution, defined based on clinical presentation, clinical course (showing a progressive deterioration of conscious within the first 24-48 h), and neuroradiological findings.
* Age: ≥ 18 years at admission
* Informed consent of the patient or consent of patient's next of kin (plus consent of an independent physician)

Exclusion Criteria:

* Patients with wounds, scars including the front orbital region.
* Patients with any known ocular condition that may be worsened by sustained eye pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Increased intracranial pressure | 24 months
  The primary outcome is the non-invasive, absolute intra-cranial pressure (ICP) in M-MCA patients before decompressive surgery, as determined by the "non-invasive ICP absolute value meter" in mmHg

SECONDARY OUTCOMES:
Correlation of ICP, neuroimaging and transcranial color Doppler | 24 months
  Correlation between non-invasive measured ICP and clinical and neuroimaging findings and standard transcranial color Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Javier Fandino, Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau AG, Aarau, Switzerland